CLINICAL TRIAL: NCT02192892
Title: Acceptability of α-amylase Fortified Blended Foods Among Children 12-36 Months Old Children and Caregivers in Burkina Faso
Brief Title: Acceptability Among Children and Caregivers of Amylase Porridges
Acronym: AMY-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Food Specialties (Industry)
Collaborators: United Nations World Food Programme (WFP) (Other)
Responsible Party: Principal Investigator, Van Hoan Nguyen, Program Officer, United Nations World Food Programme (WFP)
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 2013-10-28-AmyVisc
Record Dates: First submitted 2014-06-12; First posted 2014-07-17 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Malnutrition
Keywords: Young children; Acceptability; Food intake; Energy dense porridge
MeSH Terms: conditions — Malnutrition | interventions — Placental Lactogen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (18):
- CSB drum dried + α-amylase (Experimental): CSB drum dried + α-amylase: Porridge from Corn Soy Blend drum dried with α-amylase
  Interventions: Dietary Supplement: CSB drum dried + α-amylase
- CSB drum dried - α-amylase (Placebo Comparator): CSB drum dried - α-amylase: Porridge from Corn Soy Blend drum dried without α-amylase
  Interventions: Dietary Supplement: CSB drum dried + α-amylase
- CSB + α-amylase (Experimental): CSB + α-amylase: Porridge from Corn Soy Blend with α-amylase
  Interventions: Dietary Supplement: CSB + α-amylase
- CSB - α-amylase (Placebo Comparator): CSB - α-amylase: Porridge from Corn Soy Blend without α-amylase
  Interventions: Dietary Supplement: CSB + α-amylase
- RSB + α-amylase (Experimental): RSB + α-amylase: Porridge from Rice Soy Blend with α-amylase
  Interventions: Dietary Supplement: RSB + α-amylase
- RSB - α-amylase (Placebo Comparator): RSB - α-amylase: Porridge from Rice Soy Blend without α-amylase
  Interventions: Dietary Supplement: RSB + α-amylase
- WSB + α-amylase (Active Comparator): WSB + α-amylase: Porridge from Wheat Soy Blend with α-amylase
  Interventions: Dietary Supplement: WSB + α-amylase
- Commercial porridge flour (Active Comparator): Porridge from commercial porridge flour
  Interventions: Dietary Supplement: Commercial porridge flour
- Commercial porridge bar (Active Comparator): Porridge from commercial porridge bar
  Interventions: Dietary Supplement: Commercial porridge bar
- CSB PLUS drum dried + α-amylase (Experimental): CSB PLUS drum dried + α-amylase: Porridge from Corn Soy Blend PLUS drum dried with α-amylase
  Interventions: Dietary Supplement: CSB PLUS drum dried + α-amylase
- CSB PLUS drum dried - α-amylase (Placebo Comparator): CSB PLUS drum dried - α-amylase: Porridge from Corn Soy Blend PLUS drum dried without α-amylase
  Interventions: Dietary Supplement: CSB PLUS drum dried + α-amylase
- CSB PLUS + α-amylase (Experimental): CSB PLUS + α-amylase: Porridge from Corn Soy Blend PLUS with α-amylase
  Interventions: Dietary Supplement: CSB PLUS + α-amylase
- CSB PLUS - α-amylase (Placebo Comparator): CSB PLUS - α-amylase: Porridge from Corn Soy Blend PLUS without α-amylase
  Interventions: Dietary Supplement: CSB PLUS + α-amylase
- RSB PLUS + α-amylase (Experimental): RSB PLUS + α-amylase: Porridge from Rice Soy Blend PLUS with α-amylase
  Interventions: Dietary Supplement: RSB PLUS + α-amylase
- RSB PLUS - α-amylase (Placebo Comparator): RSB PLUS - α-amylase: Porridge from Rice Soy Blend PLUS without α-amylase
  Interventions: Dietary Supplement: RSB PLUS + α-amylase
- WSB PLUS + α-amylase (Experimental): WSB PLUS + α-amylase: Porridge from Wheat Soy Blend PLUS with α-amylase
  Interventions: Dietary Supplement: WSB PLUS + α-amylase
- WSB PLUS - α-amylase (Placebo Comparator): WSB PLUS - α-amylase: Porridge from Wheat Soy Blend PLUS without α-amylase
  Interventions: Dietary Supplement: WSB PLUS + α-amylase
- Commercial MSB + α-amylase (Active Comparator): Commercial MSB + α-amylase: Commercial porridge from Mais Soy Blend with α-amylase
  Interventions: Dietary Supplement: Commercial MSB + α-amylase

INTERVENTIONS:
Dietary Supplement: CSB drum dried + α-amylase — CSB drum dried + α-amylase: Porridge from drum dried Corn Soy Blend with α-amylase
  Arms: CSB drum dried + α-amylase; CSB drum dried - α-amylase
Dietary Supplement: CSB + α-amylase — CSB + α-amylase: porridge from Corn Soy Blend with α-amylase
  Arms: CSB + α-amylase; CSB - α-amylase
Dietary Supplement: RSB + α-amylase — RSB + α-amylase: Porridge from Rice Soy Blend with α-amylase
  Arms: RSB + α-amylase; RSB - α-amylase
Dietary Supplement: WSB + α-amylase — WSB + α-amylase: Porridge from Wheat Soy Blend with α-amylase
  Arms: WSB + α-amylase
Dietary Supplement: CSB PLUS drum dried + α-amylase — CSB PLUS drum dried + α-amylase: Porridge from drum dried Corn Soy Blend PLUS with α-amylase
  Arms: CSB PLUS drum dried + α-amylase; CSB PLUS drum dried - α-amylase
Dietary Supplement: CSB PLUS + α-amylase — CSB PLUS + α-amylase: Porridge from Corn Soy Blend PLUS with α-amylase
  Arms: CSB PLUS + α-amylase; CSB PLUS - α-amylase
Dietary Supplement: RSB PLUS + α-amylase — RSB PLUS + α-amylase: Porridge from Rice Soy Blend PLUS with α-amylase
  Arms: RSB PLUS + α-amylase; RSB PLUS - α-amylase
Dietary Supplement: WSB PLUS + α-amylase — WSB PLUS + α-amylase: Porridge from Wheat Soy Blend PLUS with α-amylase
  Arms: WSB PLUS + α-amylase; WSB PLUS - α-amylase
Dietary Supplement: Commercial porridge flour — Porridge from commercial porridge flour
  Arms: Commercial porridge flour
Dietary Supplement: Commercial porridge bar — Porridge from commercial porridge bar
  Arms: Commercial porridge bar
Dietary Supplement: Commercial MSB + α-amylase — Commercial MSB + α-amylase: Commercial porridge from Mais Soy Blend with α-amylase
  Arms: Commercial MSB + α-amylase

SUMMARY:
Addition of α-amylase is considered as one of most effective solution to improve energy density of cereal based porridges (WHO, 2008). By adding α-amylase, the viscosity of porridges will be decreased while keeping dry matter content constant. Potential positive impact is to significantly improve efficiency of WFP nutritional programmes targeting vulnerable groups suffering from acute malnutrition.

The acceptance of porridges made with α-amylase is tested compared to porridges made without α-amylase among 12-36 months old children and their caregivers. Acceptance is measured based on energy intake. The porridges tested consist of fortified blended Supercereal (12- <24 months) and Supercereal-Plus (24-36 months) based on Corn Soy Blend (CSB) extruded or drum dried, Wheat Soy Blend (WSB), Rice Soy Blend (RSB), all with and without α-amylase, or a commercial porridge, or eeZee bar.

DETAILED DESCRIPTION:
In total 120 caregiver-child pairs will be recruited in in a rural area in Fada N'Gourma Province, Burkina Faso. In total 240 subjects are included in the study: 80 children aged 12-23.9 months with 80 caregivers and 40 children aged 24-36 months with 40 caregivers. Per group (12-23.9 months or 24-36 months) 10 porridges will be prepare according to cooking instructions at central points of the villages where children are living. The caregiver will feed porridge to their children. Children eat as much porridge as they like. Porridge energy, micro- and macronutrient intake will be determined and porridge viscosity. Children and caregivers are randomly assigned to 10 different porridges, one meal per day and 3 consecutive days per porridge. Total duration is consecutively 30 days. The 120 caregivers will participate in a sensory test. At the end of the study, all caregivers will evaluate sensory of 5 out of the 10 porridges by survey, by ranking and by interview.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12 to 36 months
* Anthropometry (for children only): MUAC > 115 mm
* Informed signed consent of parents/caregivers
* Beside breastfeeding, children are used to consume complementary foods

Exclusion Criteria:

* Illness or any medical complications at the recruitment time
* Children already enrolled in any Feeding Program

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Energy intake by children | 1 day
  Energy intake (kcal/d) by children calculated on the basis of actual intake of wet weight porridge and converted into dry weight (grams). Mean of three measures on three different days.

SECONDARY OUTCOMES:
Viscosity of porridge | 1 day
  Viscosity by Bostwick consistometer (cm/30 secs). Mean of three measures on three different days.
Micronutrient and macronutrient intake by children | 1 day
  Micronutrient and macronutrient intake (mg/d) children calculated on the basis of actual intake of wet weight porridge and converted into dry weight (grams). Mean of three measures on three different days.
Acceptability of porridge by caregivers | 1 day
  Acceptability of caregivers ("liking" on a 5-point Hedonic scale, by ranking and by interview)

CONTACTS AND LOCATIONS:
Locations (1):
- GRET, Fada N'gourma, Fada N'Gourma Province, Burkina Faso

REFERENCES:
- [Derived] Kampstra NA, Van Hoan N, Koenders DJPC, Schoop R, Broersen BC, Mouquet-Rivier C, Traore T, Bruins MJ, de Pee S. Energy and nutrient intake increased by 47-67% when amylase was added to fortified blended foods-a study among 12- to 35-month-old Burkinabe children. Matern Child Nutr. 2018 Jan;14(1):e12459. doi: 10.1111/mcn.12459. Epub 2017 May 3. PMID 28466569